CLINICAL TRIAL: NCT02036203
Title: A Prospective, Randomized, Single Blind, Two Arms Controlled Study of the Safety and Efficacy of the SCu300A IUB™ Spherical Copper Intrauterine Ball in Comparison to TCu 380 IUD Intra-uterine Contraceptive Device
Brief Title: A Study on the Safety and Efficacy of the SCu300A IUB Compared to the TCu380 Copper IUD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn prior to patients enrolment due to sponsor's decision
Sponsor: Ocon Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AOS-2000-05
Record Dates: First submitted 2013-12-23; First posted 2014-01-14 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Reversible Prevention of Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCu300A IUB (Experimental)
  Interventions: Device: SCu300A IUB
- TCu380A (Active Comparator)
  Interventions: Device: TCu380A IUD

INTERVENTIONS:
Device: SCu300A IUB — Spherical copper contraceptive
  Arms: SCu300A IUB
Device: TCu380A IUD — T-shaped copper IUD
  Arms: TCu380A

SUMMARY:
This study aims to evaluate the safety and efficacy of the IUB SCu300A spherical copper IUD compared to the standard T shaped copper IUD, the TCu380.

Participants will be followed for one year and quality of life measurements will be measured during this period as well.

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 25-42

* Free and willing to fully comply with treatment process
* Healthy women seeking LARC
* Married or in a steady relationship (at least 1 year)
* Blood hemoglobin >11.5gr%
* Signed informed consent form
* If took COCP at least had one cycle after use of OC

Exclusion Criteria(major)

* Use IUB/IUD as an emergency contraception
* A previously placed IUD that has not been removed
* Pregnancy or suspicion of pregnancy
* Use of other contraception method (condom for either male or female, oral contraceptives, diaphragms, spermicides, hormonal patches, injections or ring, cervical cap)
* History of pelvic inflammatory disease, recent or remote.
* Postpartum endometritis or post abortal endometritis in the past 3 month
* Mucopurulent cervicitis
* Endometrial thickness more than 12 mm on insertion date
* Known anemia
* History of previous IUD complications
* Dysfunctional uterine bleeding
* Undiagnosed uterine bleeding
* Malignancy or suspected malignant disease of female inner or outer genitalia
* Distortions of the uterine cavity by uterine fibroids or known anatomical abnormalities
* Known intolerance or allergy to nitinol or copper and/or copper IUDs - Wilson's disease.
* Medication that may interfere with the subject's ability to complete the protocol
* Use of injectable contraception in the previous year
* Any other significant disease or condition that could interfere with the subject's ability to complete the protocol
* A history of alcohol or drug abuse
* Known infection with human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Pregnancy or pregnancy planned during the year
* Enrollment (less than 30 days after completing another study) in or planned to be enrolled in another study

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2014-01-14 (Actual); Study Completion 2014-01-14 (Actual)

PRIMARY OUTCOMES:
Perforation rate | During device insertion
  Number of subjects with partial or complete perforation through the uterine wall
Device expulsion | 12 months
  Number of subjects with partially or fully ejected devices
Efficacy in preventing pregnancy | 12 months
  Number of women who become pregnant during the trial period.
Device malposition | 12 months
  Number of subjects with observed device malposition within the uterine cavity

SECONDARY OUTCOMES:
Menorrhagia and dysmenorrhea rates | 12 months
  Recording of menstrual pain, cramps and irregular bleeding as reported by subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Center, Netanya, Israel